CLINICAL TRIAL: NCT00003338
Title: The Utility of LymphoScan Imaging in the Dectection of Residual Tumor After Chemotherapy and/or Radiotherapy in Patients With Non-Hodgkin's Lymphoma
Brief Title: Monoclonal Antibodies in Detecting Residual Disease in Patients Who Have Been Treated for Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Purpose: Diagnostic
Other Study IDs: CDR0000066309; IM-D-LL2-06; NCI-V98-1418
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2001-12

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Radioimmunodetection; epratuzumab

INTERVENTIONS:
Procedure: immunoscintigraphy
Radiation: technetium Tc 99m epratuzumab

SUMMARY:
RATIONALE: Diagnostic imaging procedures, such as radiolabeled monoclonal antibodies, may improve the ability to detect the residual disease in patients who have been treated for non-Hodgkin's lymphoma.

PURPOSE: Phase II/III trial to study the effectiveness of monoclonal antibodies in detecting residual disease in patients who have been treated for non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety of multiple (2-3) administrations of technetium Tc 99m LL2 monoclonal antibody (LymphoScan) in patients with B-cell non-Hodgkin's lymphoma after chemotherapy and/or radiotherapy. II. Describe human antimouse antibody production in these patients. III. Demonstrate that addition of a single LymphoScan study to conventional diagnostic modalities (CDMs) can differentiate between tumor and residual scarring. IV. Determine the diagnostic operating characteristics of LymphoScan to detect residual tumor in patients with radiologically detectable masses. V. Compare patient management plans based on CDMs alone and both CDMs and LymphoScan.

OUTLINE: This is an open label, multicenter study. Patients receive an infusion of technetium Tc 99m LL2 monoclonal antibody (LymphoScan) by IV injection or infused over 20-30 minutes after completion of therapy as part of the response evaluation procedures. Planar images are acquired between 4-8 hours and 18-24 hours following antibody injection, and single photon emission computerized tomography (SPECT) imaging is performed between 4-8 hours following antibody injection. Patients may receive a repeat injection of LymphoScan. Patients are followed for 3 to 6 months.

PROJECTED ACCRUAL: There will be 60 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed B-cell non-Hodgkin's lymphoma (low, intermediate, or high grade categories) Must have been treated with chemotherapy and/or radiotherapy with evidence of minimal residual disease by conventional diagnostic modalities A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: BUN no greater than 1.5 times upper limit of normal (ULN) Creatinine no greater than 1.5 times ULN Other: No known allergies to mouse proteins No second primary malignancy within past 5 years other than adequately treated in situ carcinoma of the cervix or uterus, or basal or squamous cell carcinoma of the skin Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior exposure to mouse antibodies other than LymphoScan Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified Other: At least 1 month since any other prior investigational therapy No concurrent participation in another protocol involving medical devices or investigational agents

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: William A. Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (8):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Nuclear Physicians Ltd., Cuyahoga Falls, Ohio
  - University of Texas- Houston Medical School, Houston, Texas
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Istituto Europeo Di Oncologia, Milan, Italy
- Lund University Hospital, Lund, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland